CLINICAL TRIAL: NCT06907069
Title: A Multicenter, Prospective, Open-label Clinical Study on the Treatment of Carbapenem Resistant Gram-negative Bacterial Lung Infection With Sodium Polycolistin E Mesylate Intravenically Combined With Atomization
Brief Title: Polycolistin E Sodium Mesylate Combined With Intravenous Atomization for Carbapenem Resistant Gram-negative Bacteria in Pulmonary Infection
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-R044-02
Record Dates: First submitted 2024-12-09; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lung Infection Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenously atomized polycolistin E sodium mesylate (Experimental)
  Interventions: Drug: Intravenously atomized polycolistin E sodium mesylate

INTERVENTIONS:
Drug: Intravenously atomized polycolistin E sodium mesylate — To explore the therapeutic effect of CMS combined with intravenous atomization in patients with carbapenem resistant gram-negative bacteria in lung infection.

SUMMARY:
Pulmonary infection is a kind of infectious disease that seriously damages human health. It usually starts quickly and progresses rapidly in clinical manifestations, and is often accompanied by upper respiratory tract infection symptoms. With the increasing use of broad-spectrum antibiotics in clinical practice, the failure of anti-infection caused by drug-resistant bacteria is more and more common. Once a patient develops carbapenem-resistant gram-negative bacteria (CRO) infection, there are limited drug options. Therefore, HAP, as a serious and common complication, has a high incidence and mortality for ICU patients. In this study, patients who met the diagnostic criteria for pulmonary infection caused by CRO that was clearly or strongly suspected to be resistant to carbapenems but sensitive to CMS were selected, and the combined treatment regimen of CMS intravenous atomization was adopted. To explore the therapeutic effect of CMS combined with intravenous atomization in patients with carbapenem resistant gram-negative bacteria in lung infection. To evaluate the safety and tolerability of the combination regimen in patients with pulmonary infections caused by CRO. The purpose of this study was to explore the efficacy and safety of CMS combined with intravenous atomization in the treatment of patients with CRO induced pulmonary infection, and to provide a basis for its clinical rational application.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent;
2. Inpatients aged 18-80 years old, regardless of gender;
3. Patients who met the diagnostic criteria for pulmonary infection in the Guidelines for the Diagnosis and Treatment of Hospital-Acquired Pneumonia and Ventilator-Associated Pneumonia for Adults in China (2018 Edition);
4. Infections caused by Gram-negative bacteria (CRO) that are known or strongly suspected to be resistant to carbapenems but sensitive to CMS.

Exclusion Criteria:

1. Age > 80 years old;
2. The patient had a history of severe allergy or hypersensitivity to polymyxins;
3. Patients with serious dysfunction of heart, liver, kidney and other important organs;
4. Patients with serious diseases such as malignant tumors and blood system diseases;
5. Patients with low immune function and risk of opportunistic pathogen infection;
6. Patients who used excessive colistin intravenous or atomized inhalation therapy within 72h before enrollment;
7. Have participated in other clinical trials within three months;
8. Pregnant or breastfeeding women;
9. There are other circumstances that the researcher believes are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical effective rate | From enrollment to the end of treatment at 14 days
  Clinical effective rate = (number of effective cases/total number of treated cases) × 100% Effective cases are those that include complete response (disappearance of symptoms), partial response (significant improvement in symptoms), or those that meet specific efficacy criteria.
  Inactive cases are patients whose symptoms do not improve or worsen.

SECONDARY OUTCOMES:
Microbial clearance | 14-day treatment
  The microbial clearance rate can be calculated by calculating the change in the number of microorganisms before and after disinfection. Specifically, the number of microorganisms before disinfection minus the number of microorganisms after disinfection, divided by the number of microorganisms before disinfection, to obtain the proportion of microbial reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Z, China